CLINICAL TRIAL: NCT00629928
Title: A Comparative Efficacy and Safety of Nexium Delayed-Release Capsules (40mg qd and 20mg qd) Versus Placebo for the Prevention of Gastric and Duodenal Ulcers Associated With Daily NSAID Use in Patients at Risk
Brief Title: Ulcer Prevention II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SH-NEN-0014; D9617C00014
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: NSAID Associated Gastric Ulcers
Keywords: NSAID, Nexium, esomeprazole, Gastric Ulcers
MeSH Terms: conditions — Stomach Ulcer | interventions — Esomeprazole

ARMS (3):
- 1 (Experimental): 20mg capsule once daily
  Interventions: Drug: Esomeprazole
- 2 (Experimental): 40mg capsule daily
  Interventions: Drug: Esomeprazole
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 20mg oral capsule daily
  Other Names: Nexium
  Arms: 1
Drug: Esomeprazole — 40mg oral capsule daily
  Other Names: Nexium
  Arms: 2
Drug: Placebo
  Arms: 3

SUMMARY:
Nonsteroidal anti-inflammatory drugs (NSAIDS) are often associated with gastric ulcers. This study looks at the prevention of these gastric ulcers, in patients deemed to be at risk, with either esomeprazole 40 mg once daily; esomeprazole 20 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

1. No active/current gastric or duodenal ulcer on baseline endoscopy.
2. A clinical diagnosis of a chronic condition that requires daily NSAID treatment for at least 6 months.
3. Other inclusion criteria, as defined in the protocol.

Exclusion Criteria:

1. History of esophageal, gastric or duodenal surgery, except the simple closure of an ulcer.

* 2. History of severe liver disease, including (but not limited to) cirrhosis and acute or chronic hepatitis.
* 3. Other criteria, as defined in the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2001-02; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of esomeprazole 40 mg qd versus placebo and esomeprazole 20 mg qd versus placebo for up to 6 months of treatment for the prevention of gastric (and duodenal) ulcers in patients receiving daily NSAID therapy. | Assessments at Week 0, Week 4, Week 12, Week 26

SECONDARY OUTCOMES:
Investigator assessed symptoms, defined as control of NSAID-associated GI symptoms for up to 6 months of treatment with esomeprazole 40 mg qd versus placebo and esomeprazole 20 mg qd versus placebo in patients receiving daily NSAID therapy. | Assessments at Week 0, Week 4, Week 12, Week 26
Safety and tolerability of esomeprazole 40 mg qd versus placebo and esomeprazole 20 mg qd versus placebo when administered for up to 6 months to patients receiving daily NSAID therapy. | Assessments at Week 0, Week 4, Week 12, Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca